CLINICAL TRIAL: NCT01822483
Title: A Prospective Study to Investigate Mycophenolic Acid (MPA) Exposure Through Area Under the Curve (AUC) in Renal Transplants Recipients Treated With Mycophenolate Mofetil (MMF) and After Conversion to Mycophenolate Sodium (EC-MPS)
Acronym: AUC-MPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Valter Duro Garcia, PHYSICIAN NEPHROLOGY, Irmandade Santa Casa de Misericórdia de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CERL080; CERL080ABR08T (Other: NOVARTIS)
Record Dates: First submitted 2013-03-21; First posted 2013-04-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation; mycophenolic acid; mycophenolate mofetil; mycophenolate sodium; area under the curve
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate sodium (Experimental): Arm1(Conversion):MPA AUC below 30mcg*h ml-1 - MPS+Calcineurin inhibitor+prednisone
  Interventions: Drug: Mycophenolate sodium
- Mycophenolate mofetil (Active Comparator): Arm2(Maintained):MPA AUC between 30 to 60 mg*h ml-1 or above 60 mg - MMF+Calcineurin inhibitor+prednisone
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate sodium — The conversion will be performed abruptly for all patients. Mycophenolate mofetil will be discontinued one day before the day of conversion (Day 1). Mycophenolate sodium will be introduced on day 1 with equivalent doses.
  Arms: Mycophenolate sodium
Drug: Mycophenolate mofetil — Mycophenolate mofetil dose will be maintained or adjusted to keep 30 to 60 mg*h ml-1.
  Arms: Mycophenolate mofetil

SUMMARY:
The purpose of this study is investigate mycophenolic acid exposure through area under the curve in renal transplants recipients treated with mycophenolate mofetil and after conversion to mycophenolate sodium.

DETAILED DESCRIPTION:
A growing body of evidence has shown that mycophenolate acid (MPA) exposure assessment and dosage adjustment are necessary in patients treated with mycophenolate mofetil (MMF), but there is still limited information about the dose-exposure-effect relationship of the enteric-coated mycophenolate sodium (EC-MPS) formulation that has quite different physicochemical properties (TETT et al., 2011).

Pharmacokinetically guided exposure-controlled area under the concentration-time curve (AUC) approaches are helpful to limit interpatient variability of MPA exposure and to improve the clinical outcome of organ transplant recipients (TETT et al., 2011).

MPA area under the concentration-time curve values between 30 and 60 μg h/mL in the early post-transplant period reduces the risk of acute rejections and seems to be appropriate in renal allograft recipients taking mycophenolate sodium (MPS) and calcineurin inhibitors (GRINYÓ et al., 2009; SOMMERER et al., 2010).

Among the benefits of therapeutic drug monitoring of MPA are the evaluation of interaction between MPA and proton pump inhibitors and association of donor-specific antibodies reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening;
* Subjects above the sixth month post renal transplant;
* Subjects receiving mycophenolate mofetil;
* Women of childbearing potential (CBP) with a negative pregnancy test at screening (urine or serum);
* Women of CBP and men with sexual partners of CBP must agree to use a medically acceptable method of contraception throughout the study.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, are not able to complete the study;
* Recipients of multiple organ transplant (i.e., prior or concurrent transplantation of a non-renal allograft;
* Use of any investigational drug or treatment up to 4 weeks before enrollment;
* Subjects with a calculated GFR < 30ml/min (abbreviated MDRD formula);
* Subjects with a screening total white blood cell count (WBC) ≤ 2000/mm3, hemoglobin ≤ 10g/dL and platelet count ≤ 100000/mm3;
* TGO/AST, TGP/ALT and bilirubin with values three times higher that reference values;
* History of malignancy within 3 years enrollment other than adequately treated basal cell or squamous cell carcinoma of the skin;
* Subjects who are known to be human immunodeficiency virus (HIV), hepatitis B or hepatitis C;
* Chronic hepatic failure;
* Planned treatment with immunosuppressive therapies other than those described in the protocol;
* Recipients who required desensitization protocols.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the frequency of renal transplants recipients taking mycophenolate mofetil (MMF) with MPA AUC below target level (30mcg*h ml-1). | Baseline
  Evaluate the frequency of renal transplants recipients taking mycophenolate mofetil (MMF) with MPA AUC below target level (30mcg*h ml-1).

SECONDARY OUTCOMES:
Evaluate the association of MPA AUC in renal transplant recipients with donor specific antibodies (DSA); | Baseline; month 6.
  Evaluate the association of MPA AUC in renal transplant recipients with donor specific antibodies (DSA);
Evaluate the interaction between MMF or EC-MPS and the proton pump inhibitor omeprazole through the AUC in patients with MPA below target level (30mcg*h ml-1). | 6 months
  Evaluate the interaction between MMF or EC-MPS and the proton pump inhibitor omeprazole through the AUC in patients with MPA below target level (30mcg*h ml-1).
Evaluate the association of MPA AUC with renal function estimated by MDRD formula. | Baseline; day one; months 2, 4 and 6.
  Evaluate the association of MPA AUC with renal function estimated by MDRD formula.
Evaluate the MPA_AUC in renal transplant patients converted to mycophenolate sodium (MPS) with equivalent dose of mycophenolate mofetil (MMF). | Baseline, five days after day one, fourteen days after day one, months 2,4 and 6
  Evaluate the MPA_AUC in renal transplant patients who were taking mycophenolate mofetil (MMF) and were converted to the use of mycophenolate sodium (MPS) by having the MPA concentration below the target level of 30 mcg*h ml-1.
Evaluate the MPA_AUC in renal transplant patients maintained with mycophenolate mofetil (MMF). | baseline, months 2,4 and 6
  Evaluate the AUC_MPA in renal transplant patients maintained with mycophenolate mofetil(MMF) by having the MPA concentration between 30-60 mcg*h ml-1

CONTACTS AND LOCATIONS:
Overall Officials: Valter Garcia, Physician, Principal Investigator — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Elizete Keitel, Physician, Study Chair — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Daniela Seelig, Physician, Study Chair — IRMANDADE DA SANTA CASA DE MISERICÓRIDA DE PORTO ALEGRE; Fabiano Klaus, Physician, Study Chair — IRMANDADE DA SANTA CASA DE MISERICÓRIDA DE PORTO ALEGRE; Ronivan Dal Pra, Pharmacist, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Larissa Pacheco, Pharmacist, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Bruna Cardoso, Pharmacist, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Roger Kist, Trainee, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE; Helen Zanetti, Pharmacist, Study Director — IRMANDADE DA SANTA CASA DE MISERICÓRDIA DE PORTO ALEGRE
Locations (1):
- Irmandade Da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Tett SE, Saint-Marcoux F, Staatz CE, Brunet M, Vinks AA, Miura M, Marquet P, Kuypers DR, van Gelder T, Cattaneo D. Mycophenolate, clinical pharmacokinetics, formulations, and methods for assessing drug exposure. Transplant Rev (Orlando). 2011 Apr;25(2):47-57. doi: 10.1016/j.trre.2010.06.001. Epub 2010 Dec 28. PMID 21190834
- [Background] Grinyo JM, Ekberg H, Mamelok RD, Oppenheimer F, Sanchez-Plumed J, Gentil MA, Hernandez D, Kuypers DR, Brunet M. The pharmacokinetics of mycophenolate mofetil in renal transplant recipients receiving standard-dose or low-dose cyclosporine, low-dose tacrolimus or low-dose sirolimus: the Symphony pharmacokinetic substudy. Nephrol Dial Transplant. 2009 Jul;24(7):2269-76. doi: 10.1093/ndt/gfp162. Epub 2009 Apr 8. PMID 19357111
- [Background] Sommerer C, Muller-Krebs S, Schaier M, Glander P, Budde K, Schwenger V, Mikus G, Zeier M. Pharmacokinetic and pharmacodynamic analysis of enteric-coated mycophenolate sodium: limited sampling strategies and clinical outcome in renal transplant patients. Br J Clin Pharmacol. 2010 Apr;69(4):346-57. doi: 10.1111/j.1365-2125.2009.03612.x. PMID 20406219